CLINICAL TRIAL: NCT07215754
Title: Real World Evidence of Anifrolumab in Systemic Lupus Erythematosus: a Multicenter Spontaneous Observational Study Aimed at Evaluating the Efficacy and Safety of Anifrolumab in a Cohort of Patients With Active Systemic Lupus Erythematosus
Brief Title: Real World Evidence of Anifrolumab in Systemic Lupus Erythematosus: Investigator Initiated, Observational, Multicenter Study Evaluating Effectiveness and Safety of Anifrolumab in Active SLE Patients
Acronym: REVEAL
Status: Recruiting | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Marta Mosca, Full Professor of Rheumatology, University of Pisa
Other Study IDs: 24198
Record Dates: First submitted 2025-10-02; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; Anifrolumab; Real World Evidence
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BACKGROUND AND RATIONALE. The role of type I interferons (IFN) in innate and adaptive immunity has been extensively studied, establishing a key role for type I IFNs in immune homeostasis. With growing evidence that type I IFNs play an important role in autoimmune diseases, inhibition of type I IFN biological activity with Anifrolumab represents a significant therapeutic option in SLE. Phase II and III clinical trials have demonstrated the efficacy and safety of the drug in patients with moderate-to-severe active disease.

OBJECTIVES. The primary objective of the study is to evaluate the clinical efficacy and incidence of adverse events associated with Anifrolumab therapy in a multicenter cohort of patients with SLE. Secondary objectives of the study are: - to evaluate the efficacy of therapy on different types of clinical manifestations; - to assess the impact of therapy on quality of life and other patient-reported outcome measures (PROMs); - to evaluate the steroid-sparing potential of therapy; - to assess the speed of therapeutic action on different clinical manifestations; - to identify predictive variables of clinical response to therapy; - to evaluate drug retention rate; - to assess the efficacy of therapy in reducing organ damage accumulation.

PRIMARY AND SECONDARY ENDPOINTS. Primary efficacy endpoints: - Percentage of patients in remission (DORIS criteria) at 6, 12, 24, 36, 48, and 60 months; - Percentage of patients in low disease activity state (LLDAS) at 6, 12, 24, 36, 48, and 60 months. Secondary efficacy endpoints: - Incidence of disease flares according to the modified SFI; - Percentage of patients with organ damage accumulation (SLICC/DI > 0) compared to baseline at 12, 24, 36, 48, and 60 months; - Longitudinal changes in disease activity indices SLEDAI-2K and SLE-DAS; - Percentage of patients on steroid therapy ≤5 mg prednisone equivalent and percentage of patients who discontinued steroids at 6, 12, 24, 36, 48, and 60 months; - Longitudinal changes in PROMs (quality of life, fatigue, pain, PGA); - Longitudinal changes in Physician's Global Assessment and Patient's Global Assessment; - Longitudinal changes in CLASI score (in patients with cutaneous manifestations); - Longitudinal changes in joint count (in patients with articular manifestations); - Evaluation of predictive variables of response to therapy; - Evaluation of "time to response". Primary safety endpoints: - Incidence of adverse events (serious and non-serious). Secondary safety endpoints: - Incidence of serious adverse events; - Incidence of hospitalizations due to adverse events; - Incidence of infections (particularly Herpes Zoster and its outcomes); - Incidence of cardiovascular events; - Incidence of neoplasms or precancerous lesions.

ELIGIBILITY. Inclusion criteria: - Patients diagnosed with SLE according to classification criteria valid at diagnosis time (1997, 2012, 2019); - Written informed consent; - Active disease for which the patient is a candidate for Anifrolumab treatment (including compassionate use); - Active disease for which the patient has started Anifrolumab treatment. Exclusion criteria: - Age <18 years; - Absence of patient consent. Withdrawal criteria: - Patient withdrawal of consent.

STUDY TIMELINES. Duration per patient: 60 months. Enrollment period: 3 years. Total study duration: 5 years.

SAMPLE SIZE CALCULATION. Due to the study design and novelty of the topic, a formal sample size calculation is not feasible. However, based on disease frequency, estimated flare rates over one year, and the number of centers involved, at least 150 patients are expected to be enrolled. The study population will be analyzed by intention-to-treat (ITT), including all enrolled patients. For the primary safety and efficacy endpoints, the percentage of patients in remission and low disease activity, as well as event incidence, will be calculated over 60 months. An interim analysis is planned when the first 50 patients complete the 24-week evaluation. Adverse event incidence will be summarized overall, by severity (SAE, any AE), time of onset (early, late), and relationship to the study treatment. Disease flare incidence will be summarized overall and by severity. Time-to-event for disease occurrence will be evaluated using Kaplan-Meier method. Analyses will be performed using STATA software, with statistical significance set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with SLE according to classification criteria valid at diagnosis time (1997, 2012, 2019)
* Written informed consent
* Active disease for which the patient is a candidate for Anifrolumab treatment (including compassionate use)
* Active disease for which the patient has started Anifrolumab treatment

Exclusion Criteria:

* Age <18 years
* Absence of patient consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with SLE starting treatment with Anifrolumab according to the AIFA indications will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
attainement of remission and LLDAS | 6, 12, 24, 36, 48 and 60 months
  percentage of patients reaching the target of remission and low disease activity state

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tani C, Cardelli C, Moroni L, Zen M, Bottazzi F, Fredi M, Bortoluzzi A, Piga M, Riccio F, Ceccarelli F, De Marchi G, Manfredi L, Mule R, Biancalana E, Gatto M, Coladonato L, Conigliaro P, Gerosa M, Diamanti AP, Ramirez GA, Vesentini F, Zanframundo G, Orlandi C, Silvagni E, Chessa E, Trevisani M, Palmerini M, Pilo PFG, Ferrigno S, Di Lollo AC, Noviello S, Lo Gullo A, De Andres MI, Guiducci S, Emmi G, Maiolini F, De Angelis R, Caporali RF, Iannone F, Moroncini G, Quartuccio L, Conti F, Ciccia F, Govoni M, Franceschini F, Cavagna L, Iaccarino L, Dagna L, Mosca M. Patient profiles and early response in patients with systemic lupus erythematosus initiating anifrolumab: interim analysis from the ongoing multicentre observational REVEAL study. Lancet Rheumatol. 2026 Feb 5:S2665-9913(25)00316-9. doi: 10.1016/S2665-9913(25)00316-9. Online ahead of print. PMID 41655581